CLINICAL TRIAL: NCT04162951
Title: The Effect of Retrolaminar Thoracic Paravertebral Block on the Postoperative Analgesia of Patients Undergoing Breast Surgeries: Prospective Randomized Double Blinded Study
Brief Title: Retrolaminar Thoracic Paravertebral Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 33207/07/19
Record Dates: First submitted 2019-09-09; First posted 2019-11-14 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Regional Anesthesia Morbidity; Postoperative Pain
Keywords: Retrolaminar; Paravertebral; Breast surgery; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Prospective study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants and the investigator will be kept blinded by the aid of closed sealed envelops.
  The measurements will be collected by the aid of assistant resident who will not participating into the study and blinded to it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ordinary approach group (Experimental): The patients in this group will receive ordinary ultrasound-guided thoracic paravertebral block. by local anesthetic mixture at a volume of 0.2 ml/kg composed of plain bupivacaine 0.25% and Fentanyl 2 ug/ml.
  Interventions: Procedure: Ordinary approach paravertebral block
- Retro-laminar approach group (Experimental): The patients in this group will be receive real ultrasound-guided Retrolaminar thoracic paravertebral block by local anesthetic mixture at a volume of 0.2 ml/kg composed of plain bupivacaine 0.25% and Fentanyl 2 ug/ml.
  Interventions: Procedure: Retrolaminar paravertebral block

INTERVENTIONS:
Procedure: Ordinary approach paravertebral block — Ultrasound guided thoracic paravertebral block. At the appropriate dermatome, the needle (22-gauge, 8-10-cm, short bevelled spinal needle, or a Touhy needle if a catheter is to be placed) is inserted 2.5-3 cm lateral to the spinous process and advanced perpendicular to the skin in all planes to contact the transverse process at a variable depth (2-4 cm) depending on the build of the individual. The needle is then walked above the transverse process and gradually advanced until a loss of resistance to air or saline, or a subtle 'click' is felt as the superior costotransverse ligament is penetrated, usually within 1-1.5 cm from the superior edge of the transverse process.
  Other Names: thoracic paravvertebral blovk
  Arms: Ordinary approach group
Procedure: Retrolaminar paravertebral block — In the retrolaminar approach to TPVB or retrolaminar block (RB), local anesthetic (LA) is injected into the retrolaminar plane to achieve a truncal sensory block like that of traditional TPVB. It has been postulated that during RB, LA spreads from the injection plane to the thoracic paravertebral space (TPVS) through the superior costotransverse ligament (SCTL). Retrolaminar block will be performed under ultrasound guidance, as a single injection.
  Other Names: Thoracic retrolaminar paravertebral block
  Arms: Retro-laminar approach group

SUMMARY:
This clinical study will be conducted on female patients admitted to The General Surgery Department of Tanta Faculty of Medicine for a period of 9 months.

Patients will be randomly allocated into one of the following two groups;- • Ordinary approach group (30 patients): The patients in this group will receive ordinary ultrasound-guided thoracic paravertebral block.

• Retro-laminar approach group (30 patients): The patients in this group will be receive real ultrasound-guided Retrolaminar thoracic paravertebral block.

All the patients will receive general anesthesia with attachment to a monitor (5 ASA Monitoring) In addition to bispectral index.

DETAILED DESCRIPTION:
This prospective randomized controlled study will be carried out on female patients who will be presented for breast surgery in the General Surgery Department in Tanta university hospitals over 3 month duration and 6 months follow up that starts immediately after obtaining ethical committee approval, an informed written consent will be obtained from all the participants, all patients data will be confidential and will be used for the current study only.

Any unexpected risks that will appear during the research will be announced to the participants and to the ethical committee at time and adequate measures will be taken to resolve and avoid these risks.

Expected risks to the patients: patients enrolled in this study will have a very minimal risk of pleural puncture that will be managed by adequate observation and chest tube insertion whenever indicated. They may have a minimal risk of hypotension that will be managed by intravenous fluids and intravenous ephedrine 10 mg.

There will be adequate supervision to maintain the privacy of patients and confidentiality of data that will be used in the current study only.

There will be no conflict of interest, nor conflict with religion, law, or society standards.

The research will be beneficial to the society and has no risk of environmental pollution.

Once the patients will arrive to the operating room, intravascular access will be established, fluid preload will be started, and basic monitor will be attached. After positioning and adequate sterilization of the back. The patients will be randomly allocated into two equal groups by the aid of computer-generated software of randomization; - • Ordinary approach group (30 patients): The patients in this group will receive ordinary ultrasound-guided thoracic paravertebral block.

• Retro-laminar approach group (30 patients): The patients in this group will be receive real ultrasound-guided Retrolaminar thoracic paravertebral block.

Anesthesia will be induced by fentanyl 1.5 ug/kg, propofol 1.5 mg/kg, and cis-atracurium 0.15 mg/kg to facilitate tracheal intubation. After endotracheal intubation, the patients will be connected to a mechanical ventilator with its parameters adjusted to maintain etCo2 34-38 mmhg. Anesthesia will be maintained by isoflurane 1.5% in mixture of oxygen:air 1:1 with the use of low flow (1 ml/min).

All the patients will be connected to a bispectral index monitor with maintaining its value ranging 40-60. Increase in the BIS value over 60 will be managed by additional dose of fentanyl 1ug/kg till decrease the BIS below 60. If the BIS is still over 60, increasing the isoflurane 0.2 % MAC till it decreased below 60.

At the end of the surgery, switching off the inhalational anesthetics, reversal of muscle relaxation, and awake tracheal extubation will be done with transporting the patients to the PACU for postoperative follow up and monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Aged 40-60 years
* ASA class I-II.
* Presented for elective breast surgery.

Exclusion Criteria:

* Patients refused to participate
* Patients with known or suspected or known allergy to the used medication.
* Patients with spinal deformities.
* Patients with preoperative chronic pain,
* Patients received preoperative opioids or gabapentoids.
* Patients with major cardiac, renal, respiratory, or hepatic disease.
* Patients with suspected or diagnosed coagulopathy
* Uncooperative patients.
* Obese patients with BMI >36

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
The postoperative rescue analgesia consumption | The first 24 hours postoperatively
  Morphine consumption in the first 24 h postoperatively (3 mg morphine i.v will be given when the postoperative VAS score was 4 or more considering the total dose consumption in the first postoperative day not exceeding 15 mg.

SECONDARY OUTCOMES:
The incidence of complications | up 24 hours from performing the technique
  The incidence of complication pleural puncture, pneumothorax, hypotension, or intravascular injection .

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Ismaiel, M.D, Principal Investigator — Lecturer of Anesthesia and Intensive Care, Tanta University
Locations (1):
- Tanta University hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
Once the study had been successfully completed, the data will be shared for other researchers.